CLINICAL TRIAL: NCT02398994
Title: A Multicentre randomiSed Controlled TRial of IntraVEnous Immunoglobulin (IVIg) Versus Standard Therapy for the Treatment of Transverse Myelitis in Adults and Children
Brief Title: A Multicentre randomiSed Controlled TRial of IntraVEnous Immunoglobulin Versus Standard Therapy for Transverse Myelitis
Acronym: STRIVE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Continued effort did not successfully increase recruitment into the study.
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other); Barts and the London School of Medicine and Dentistry (Other); Cardiff University (Other); University College, London (Other); King's College Hospital NHS Trust (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Barts & The London NHS Trust (Other); Alder Hey Children's NHS Foundation Trust (Other); Walton Centre NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other); Birmingham Women's and Children's NHS Foundation Trust (Other); University Hospital Birmingham NHS Foundation Trust (Other); Cardiff and Vale University Health Board (Other Government); North Bristol NHS Trust (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Manchester University NHS Foundation Trust (Other Government); Northern Care Alliance NHS Foundation Trust (Other); University Hospital Southampton NHS Foundation Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Nottingham University Hospitals NHS Trust (Other); NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RJ115/N065; 2014-002335-34 (EudraCT Number); 11/129/148 (Other Grant/Funding Number: National Institute for Health Research, Health Technology); 12127581 (Other: ISRCTN)
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Myelitis, Transverse; Neuromyelitis Optica
Keywords: Clinical Trials Unit; Pediatric
MeSH Terms: conditions — Myelitis, Transverse; Neuromyelitis Optica | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous Methylprednisolone (Active Comparator): Paediatric patients - 30mg/kg or 500mg/m2 up to a maximum daily dose of 1g/day for 5 days.
  Adult patients - 1g/day for 5 days.
  Interventions: Drug: Intravenous Methylprednisolone
- Intravenous Immunoglobulin (Experimental): Paediatric patients <41.2kg - total dose of 2g/kg in divided doses over 2 days.
  All other patients - total dose of 2g/kg in divided doses over 5 days.
  PLUS Intravenous Methylprednisolone
  Pediatric patients - 30mg/kg or 500mg/m2 up to a maximum daily dose of 1g/day for 5 days.
  Adult patients - 1g/day for 5 days.
  Interventions: Drug: Intravenous Methylprednisolone; Drug: Intravenous Immunoglobulin

INTERVENTIONS:
Drug: Intravenous Methylprednisolone
Drug: Intravenous Immunoglobulin
  Arms: Intravenous Immunoglobulin

SUMMARY:
This multi-center randomized controlled trial evaluates if the addition of intravenous immunoglobulin to standard treatment of corticosteroids improves outcome in children and adults with first episode of Transverse Myelitis of Neuro-myelitis optica. Half of participants will receive corticosteroids alone, whilst the other half will receive corticosteroids plus intravenous immunoglobulin.

DETAILED DESCRIPTION:
Transverse myelitis (TM) is a severe demyelinating condition predominantly affecting young people, which causes significant long-term disability in approximately one third. Current initial treatment is with corticosteroids, although evidence for their use is based on extrapolation from trials in adult multiple sclerosis relapses. In view of the severity of the condition, additional treatments have been trialed.

Intravenous immunoglobulin (IVIG) is often used as second-line treatment in steroid-unresponsive central nervous system demyelination, although evidence for its efficacy is limited to small case series and case reports. Randomized controlled trials have demonstrated that IVIG reduces inflammation and enhances remyelination in a number of neurological conditions, although there have been no randomized controlled trials testing its use in adults and children with TM.

This study will evaluate if additional and early treatment with IVIG is of extra benefit in TM when compared to the current standard therapy of intravenous steroids alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of

EITHER acute first onset transverse myelitis (using the TM Consortium Working Group 2002 criteria) - patients must fulfill all of the following criteria:

* Sensory, motor, or autonomic dysfunction attributable to spinal cord disease
* Bilateral signs and/or symptoms (not necessarily symmetric)
* Sensory level (except in young children <5 years where this is difficult to evaluate)
* Lack of MRI brain criteria consistent with multiple sclerosis
* Progression to nadir between 4 h and 21 days

OR first presentation of neuromyelitis optica (using standardised criteria) - patients must fulfil both absolute criteria:

* Optic neuritis
* Acute myelitis, plus two out of three supportive criteria (as Aquaporin 4 antibody (AQP4) is often not available acutely, only the first two supportive criteria would be applied),
* Brain MRI not meeting criteria for Multiple Sclerosis (MS) at disease onset
* Spinal cord MRI with contiguous T2-weighted signal abnormality extending over three or more vertebral segments, indicating a relatively large lesion in the spinal cord
* AQP4 seropositive status

  * ASIA Impairment Score of A-C
  * Randomisation to occur no later than day 5 of steroids, and, if definitely known, within 21 days from symptom onset.
  * Give assent (8-16 years)/consent to participate in the trial

Exclusion Criteria:

* Contraindication to IVIG as stated in the summary of product characteristics (SmPC), or receiving IVIG for other reasons
* Previously known systemic autoimmune disease (e.g. systemic lupus erythematosus) or any evidence of systemic inflammation during current presentation.
* Direct infectious aetiology (e.g. varicella zoster)
* Previous episode of central nervous system (CNS) inflammatory demyelination
* Acute disseminated encephalomyelitis (ADEM)
* Other causes of myelopathy not thought to be due to myelitis (e.g. nutritional, ischaemic, tumour etc.)
* Other disease which would interfere with assessment of outcome measures
* Known pregnancy
* Circumstances which would prevent follow-up for 12 month

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
2 points or greater improvement on the American Spinal Injury Association (ASIA) Impairment scale (classified A-E) | 6 months

SECONDARY OUTCOMES:
Change in ASIA motor scale (0-100) and ASIA sensory scale (0-112) | 6 months
Change in Kurtzke's expanded disability status scale (EDSS) measured with Neurostatus scoring | 6 months
EQ-5D-Y (for patients aged 8-12 years at presentation) | 6 months
EQ-5D-5L (for patients aged 13 years or over at presentation) | 6 months
International Spinal Cord Injury (SCI) Quality of Life Basic Data Set (for patients aged 13 years or over at presentation) | 6 months
Client Service Receipt Inventory (CSRI) | 6 months

OTHER OUTCOMES:
International SCI Bladder/Bowel Data Set (for patients aged 13 years or over at presentation) | 6 months
Paediatric Quality of Life Inventory™ (PedsQL) Parent Report for Toddlers (for patients aged 2-4 years at presentation) | 6 months
Paediatric Quality of Life Inventory™(PedsQL) Parent Report for Young Children (for patients aged 5-7 years at presentation) | 6 months
International SCI Pain Basic Data Set (for patients ages 13 years or over at presentation) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ming Lim, MB, PhD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (18):
- United Kingdom (18):
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - North Bristol NHS Trust, Bristol
  - University Hospital Bristol NHS Foundation Trust, Bristol
  - Cardiff and Vale University Health Board, Cardiff
  - NHS Lothian, Edinburgh
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Walton Centre NHS Foundation Trust, Liverpool
  - Great Ormond Street Children's Hospital, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - University of London and Bart's Health NHS Trust, London
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - Newcastle-upon-Tyne Hospitals NHS Trust, Newcastle
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Trust, Oxford
  - Salford Royal NHS Foundation Trust, Salford
  - University Southampton NHS Foundation Trust, Southampton

REFERENCES:
- [Derived] Absoud M, Brex P, Ciccarelli O, Diribe O, Giovannoni G, Hellier J, Howe R, Holland R, Kelly J, McCrone P, Murphy C, Palace J, Pickles A, Pike M, Robertson N, Jacob A, Lim M. A multicentre randomiSed controlled TRial of IntraVEnous immunoglobulin compared with standard therapy for the treatment of transverse myelitis in adults and children (STRIVE). Health Technol Assess. 2017 May;21(31):1-50. doi: 10.3310/hta21310. PMID 28639937
- [Derived] Absoud M, Gadian J, Hellier J, Brex PA, Ciccarelli O, Giovannoni G, Kelly J, McCrone P, Murphy C, Palace J, Pickles A, Pike M, Robertson N, Jacob A, Lim M. Protocol for a multicentre randomiSed controlled TRial of IntraVEnous immunoglobulin versus standard therapy for the treatment of transverse myelitis in adults and children (STRIVE). BMJ Open. 2015 May 25;5(5):e008312. doi: 10.1136/bmjopen-2015-008312. PMID 26009577